CLINICAL TRIAL: NCT01026077
Title: The Savella Pregnancy Registry
Acronym: SPR
Status: Terminated | Type: Observational
Why Stopped: Per the FDA, there is no regulatory requirement to continue this registry.
Sponsor: Syneos Health (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: MLN-MD-30
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Fibromyalgia
Keywords: Savella pregnant; savella pregnancy; fibromyalgia pregnant; fibromyalgia pregnancy; pregnancy registry savella
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Fibromyalgia/prospective pregnancies: Women taking Savella during pregnancy. Register prospectively, provide verbal consent.

SUMMARY:
The Savella Pregnancy Registry is a US based registry designed to monitor pregnancies exposed to Savella (milnacipran HCI). This is an observational, exposure-registration and follow-up registry designed primarily to estimate the prevalence of major congenital anomalies, and secondarily to estimate the prevalence of recognized spontaneous abortions, stillbirths, induced abortions, minor congenital anomalies, and any serious adverse pregnancy outcomes among pregnancies exposed to Savella as well as adverse outcomes observed during the first year of life in off-springs born from these exposed pregnancies. Live offspring are followed from birth until age one. The Savella Pregnancy Registry is sponsored by AbbVie (formerly Actavis PLC, Forest Laboratories Inc., and Allergan) and managed by Syneos Health.

DETAILED DESCRIPTION:
Registry enrollment is voluntary and initiated by pregnant patients or their healthcare providers (HCP). Patient-initiated reports must be verified by the HCP. Enrollment should occur as early in pregnancy as possible, preferably before any prenatal testing has occurred; however, enrollment at any time during pregnancy is allowed. Near the estimated date of delivery, the Registry prompts the HCP to provide pregnancy outcome data. If a live birth is reported, the Registry conducts follow-up with the infant's HCP at outcome, 4 months, and 12 months of age. If a birth defect is indicated, the Registry requests additional targeted follow-up information from the HCP. Data are collected on exposure to Savella, potential confounding factors, pregnancy outcome, and pediatric outcome for all live born babies. Cases are reviewed and classified according to type of birth defects. Adverse event cases are forwarded to Allergan.

ELIGIBILITY:
Inclusion Criteria:

* Females exposed to Savella during pregnancy
* Willing to provide verbal consent
* 18 y/o, US citizen

Exclusion Criteria:

* Male
* Under 18 y/o
* Females not pregnant, not exposed to Savella

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who are exposed to Savella during pregnancy.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2009-11 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2024-10-09 (Actual)

PRIMARY OUTCOMES:
The primary objective is to estimate the prevalence of major congenital anomalies among off-springs of women exposed to Savella during pregnancy. | January 2017

SECONDARY OUTCOMES:
Estimate the prevalence of spontaneous abortions, stillbirths, induced abortions, minor congenital anomalies, and adverse pregnancy outcomes. | January 2017

CONTACTS AND LOCATIONS:
Overall Officials: Sara Ephross, PhD, Principal Investigator — Sr. Advisor, Epidemiology & Health Outcomes
Locations (1):
- Syneos Health, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study and enrollment information for healthcare providers and patients — http://www.savellapregnancyregistry.com